CLINICAL TRIAL: NCT00349414
Title: A Comparison of the Safety and Efficacy of Conventional Versus Micropulse Transscleral Diode Laser Cyclophotocoagulation in Refractory Glaucoma
Brief Title: Safety Study of Conventional Versus Micropulse Transscleral Cyclophotocoagulation in Treating End-Stage Glaucoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Paul Chew, FRCSEd,MMed, National University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSRB Reference Code: A/06/164
Record Dates: First submitted 2006-07-06; First posted 2006-07-07 (Estimated); Last update posted 2008-05-15 (Estimated); Status verified 2008-05

CONDITIONS: Advanced Glaucoma; Refractory Glaucoma
Keywords: Advanced glaucoma; Refractory glaucoma; Cyclophotocoagulation; Transscleral cyclophotocoagulation; Micropulse transscleral cyclophotocoagulation
MeSH Terms: conditions — Glaucoma

INTERVENTIONS:
Procedure: Micropulse Transscleral Cyclophotocoagulation
Procedure: Conventional Transscleral Cyclophotocoagulation

SUMMARY:
The aim of this study is to compare the safety and efficacy of conventional and micropulse transscleral diode laser in the treatment of end-stage glaucoma.

DETAILED DESCRIPTION:
End-stage glaucoma is difficult to treat, and it may sometimes be unresponsive to surgery or medications. A common treatment is the conventional transscleral cyclophotocoagulaion, but it has various side effects. This study specifically aims to compare the intraocular pressure (IOP) lowering effects and the incidence of complications such as hypotony, phthisis, sympathetic ophthalmia, surface conjunctival burns, bulbar conjunctival swelling, decompensation of corneal grafts, hyphema and vitreous hemorrhage, in conventional and the newer micropulse transscleral cyclophotocoagulation.The hypothesis is that the micropulse transscleral cyclophotocoagulation will be as good or better than the conventional transscleral cyclophotocoagulation, with less complications.

ELIGIBILITY:
Inclusion Criteria:

* · More than 21 years old

  * Advanced glaucoma refractory to maximum tolerated medical and surgical treatment
  * Visual acuity worse than 6/60
  * Poor candidates for additional filtration surgery

Exclusion Criteria:

* · Any eye surgery done within 2 months of enrolment

  * Any ocular infection or inflammation
  * Unable to give informed consent

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2006-07; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients in each group that had a 30% decrease of IOP from baseline after 6 months

SECONDARY OUTCOMES:
Number of patients with complications, such as hypotony, phthisis, sympathetic ophthalmia, surface conjunctival burns, bulbar conjunctival swelling, decompensation of corneal grafts, hyphema and vitreous hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chew, FRCSEd,MMed, Principal Investigator — National University Hospital,Ophthalmology Department
Locations (1):
- National University Hospital Singapore Department of Ophthalmology, Singapore, Singapore

REFERENCES:
- [Background] Berger JW. Thermal modelling of micropulsed diode laser retinal photocoagulation. Lasers Surg Med. 1997;20(4):409-15. doi: 10.1002/(sici)1096-9101(1997)20:43.0.co;2-u. PMID 9142680
- [Background] Ho CL, Wong EY, Chew PT. Effect of diode laser contact transscleral pars plana photocoagulation on intraocular pressure in glaucoma. Clin Exp Ophthalmol. 2002 Oct;30(5):343-7. doi: 10.1046/j.1442-9071.2002.00553.x. PMID 12213158